CLINICAL TRIAL: NCT00510302
Title: Melanoma Risk-Reduction Practices Among Melanoma Patients and Their Family Members
Brief Title: Melanoma Risk-Reduction Among Patients and Family Members
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: ID02-452
Record Dates: First submitted 2007-07-31; First posted 2007-08-02 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Melanoma
Keywords: Ultraviolet Radiation; Melanoma; Questionnaire; Survey; First Degree Relative; Interview
MeSH Terms: conditions — Melanoma | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Melanoma Risk-Reduction: Patients with melanoma, their spouses/partners, and first-degree relatives (FDRs).
  Interventions: Behavioral: Questionnaire; Behavioral: Interview

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire regarding melanoma risk-reduction.
  Other Names: Survey
Behavioral: Interview — Interview via telephone about topics related to melanoma risk-reduction.

SUMMARY:
Primary Objectives:

* To conduct semi-structured interviews with melanoma patients and family members to collect descriptive information on their UVR exposure, UVR exposure-reduction practices, melanoma early detection practices, knowledge, psychosocial variables related to melanoma risk-reduction (e.g., self-efficacy, norms, and expectations), and experiences surrounding the diagnosis of melanoma in the family. Melanoma patients and family members with children will be asked about the UVR exposure and UVR exposure-reduction practices of their children, and parental practices to reduce UVR exposure among children.
* To develop behavioral and attitudinal questionnaires based on data collected during semi-structured interviews, and evaluate the appropriateness of these questionnaires using cognitive interviewing techniques.
* To develop tailored messages aimed at promoting strategies to reduce UVR exposure (e.g., wearing protective clothing, minimizing midday UVR exposure, minimizing duration of UVR exposure, using shade and sunscreen, avoiding sun lamps, and avoiding intentional tanning) and improving adherence to surveillance and screening guidelines. Messages will be developed to correspond to responses to questionnaire items.
* To assess tailored messages for their relevance, appropriateness, attractiveness and appeal, credibility, and perceived behavioral impact among melanoma patients and their family members.

DETAILED DESCRIPTION:
Participants in Part 1 of the study will be asked to be interviewed about topics related to melanoma risk-reduction, including opinions, attitudes, beliefs, and practices related to ultraviolet radiation exposure, melanoma prevention, and melanoma detection.

Participants in Part 2 of the study will be asked to complete a written questionnaire on melanoma risk-reduction and then be interviewed to obtain feedback on how the questionnaire may be refined.

Participants in Part 3 of the study will be asked to be interviewed by telephone. Participants then will receive educational material in the form of a newsletter tailored to their interview responses. Participants then will be asked to be interviewed to obtain feedback for refining the educational material. In each part of the study, the patient/family member will receive a letter describing the study and the Consent Statement for Questionnaire and Interview Studies.

Prior to the start of the interview, the Consent Statement will be read to the patient/family member. Patients/family members may or may not choose to have the interview tape-recorded. Participants may stop the interview or questionnaire at any time and may refuse to answer any questions. At any time, the patient/family member may refuse to have the interview tape-recorded. There is no treatment associated with this study.

ELIGIBILITY:
Inclusion Criteria:

* (FDRs will include siblings and adult children.) Melanoma patients are eligible if they were diagnosed with in situ, localized, or regional melanoma after January 1, 1997.
* Melanoma patients, their spouses/partners, and their first-degree relatives (FDRs) 18 years of age or older are eligible.
* Melanoma patients, their spouses/partners, and FDRs are eligible if they can speak, read, and write English.
* Melanoma patients, their spouses/partners, and FDRs are eligible if they provide informed consent.
* Spouses/partners and FDRs of melanoma patients are eligible if the patient gives permission for them to be contacted for recruitment.
* A melanoma patient's FDR is eligible if he/she is a sibling or child of the melanoma patient.

Exclusion Criteria:

* Melanoma patients, spouses/partners of patients, and FDRs of patients are not eligible if they cannot provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with melanoma, their spouses/partners, and first-degree relatives (FDRs).
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2002-11-18 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
Information on ultraviolet radiation (UVR-E) reduction + early detection practices of melanoma patients and family members | 8 Years

SECONDARY OUTCOMES:
Development of questionnaires + tailored intervention messages on melanoma risk-reduction in a high-risk population | 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Susan Peterson, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org